CLINICAL TRIAL: NCT00474045
Title: A Randomised, Parallel-group, Open-labelled, Multinational Trial Comparing the Efficacy and Safety of Insulin Detemir (Levemir®) Versus Human Insulin (NPH Insulin), Used in Combination With Insulin Aspart as Bolus Insulin, in the Treatment of Pregnant Women With Type 1 Diabetes
Brief Title: Efficacy and Safety of Insulin Detemir Versus Neutral Protamine Hagedorn (NPH) Insulin in Pregnant Women With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1687; 2006-004861-33 (EudraCT Number)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2011-12-05 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin detemir (Experimental): Individually adjusted insulin detemir injected subcutaneously as basal insulin + individually adjusted insulin aspart injected subcutaneously as bolus insulin from randomisation (gestational week 8-12) and continued until 6 weeks after delivery. If a subject was not pregnant at randomisation, treatment was given up to a maximum of 52 weeks. For subjects who became pregnant, randomised treatment was continued until 6 weeks after delivery. Subjects who were not pregnant at 52 weeks after randomisation were withdrawn
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- Neutral Protamine Hagedorn (NPH) insulin (Active Comparator): Individually adjusted NPH insulin injected subcutaneously as basal insulin + individually adjusted insulin aspart injected subcutaneously as bolus insulin from randomisation (gestational week 8-12) and continued until 6 weeks after delivery. If a subject was not pregnant at randomisation, treatment was given up to a maximum of 52 weeks. For subjects who became pregnant, randomised treatment was continued until 6 weeks after delivery. Subjects who were not pregnant at 52 weeks after randomisation were withdrawn
  Interventions: Drug: NPH insulin; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target, dose titration, s.c. (under the skin) injection
  Arms: Insulin detemir
Drug: NPH insulin — Treat-to-target, dose titration, s.c. (under the skin) injection
  Arms: Neutral Protamine Hagedorn (NPH) insulin
Drug: insulin aspart — Treat-to-target, dose titration, s.c. (under the skin) injection

SUMMARY:
This trial is conducted in Africa, Europe, North and South America and Oceania. The aim of this trial is to compare the effect and safety on blood glucose control in pregnant women with type 1 diabetes of a modern insulin analogue (insulin detemir) and human insulin (NPH insulin) given as long-acting insulin in combination with a short-acting insulin (insulin aspart).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes treated with insulin for at least 12 months
* Planning to become pregnant and have a screening HbA1c (glycosylated haemoglobin) lesser than or equal to 9.0%, or
* Pregnant with an intrauterine singleton living foetus, 8-12 weeks pregnant when joining the trial and a HbA1c lesser than or equal to 8.0% when pregnancy is confirmed

Exclusion Criteria:

* Known or suspected hypersensitivity to the trial product(s) or related products
* Untreated hyperthyroidism or hypothyroidism
* Known or suspected abuse of alcohol or narcotics
* Cardiac problems
* Impaired kidney function
* History of severe hyperemesis gravidarum
* Treatment with in-vitro fertilisation or other medical infertility treatment
* Impaired liver function
* Uncontrolled hypertension
* Proliferative retinopathy or maculopathy requiring acute treatment
* Known to be HIV (human immunodeficiency virus) positive, Hepatitis B or Hepatitis C positive
* Any concomitant medication contraindicated in pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (86):
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Pcia de Cordoba
  - Novo Nordisk Investigational Site, Salta
- Australia (9):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Elizabeth Vale, South Australia
  - Novo Nordisk Investigational Site, Clayton
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, South Brisbane
  - Novo Nordisk Investigational Site, Subiaco
  - Novo Nordisk Investigational Site, Wollongong
- Austria (4):
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Brazil (3):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São Paulo
- Canada (9):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Edmonton
  - Novo Nordisk Investigational Site, Montreal
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Toronto
  - Novo Nordisk Investigational Site, Vancouver
  - Novo Nordisk Investigational Site, Winnipeg
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (3):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, København Ø
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (10):
  - Novo Nordisk Investigational Site, Amiens
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Bondy
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Valenciennes
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Petah Tikva, Israel
- Norway (3):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Trondheim
  - Novo Nordisk Investigational Site, Tønsberg
- Poland (8):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Olsztyn
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
  - Novo Nordisk Investigational Site, Zabrze
- Russia (5):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Tyumen
- South Africa (3):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- Spain (7):
  - Novo Nordisk Investigational Site, Alcoy
  - Novo Nordisk Investigational Site, Alicante
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- United Kingdom (14):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Mathiesen ER, Damm P, Jovanovic L, McCance DR, Thyregod C, Jensen AB, Hod M. Basal insulin analogues in diabetic pregnancy: a literature review and baseline results of a randomised, controlled trial in type 1 diabetes. Diabetes Metab Res Rev. 2011 Sep;27(6):543-51. doi: 10.1002/dmrr.1213. PMID 21557440
- [Result] Mathiesen ER, Hod M, Ivanisevic M, Duran Garcia S, Brondsted L, Jovanovic L, Damm P, McCance DR; Detemir in Pregnancy Study Group. Maternal efficacy and safety outcomes in a randomized, controlled trial comparing insulin detemir with NPH insulin in 310 pregnant women with type 1 diabetes. Diabetes Care. 2012 Oct;35(10):2012-7. doi: 10.2337/dc11-2264. Epub 2012 Jul 30. PMID 22851598
- [Result] Hod M, Mathiesen ER, Jovanovic L, McCance DR, Ivanisevic M, Duran-Garcia S, Brondsted L, Nazeri A, Damm P. A randomized trial comparing perinatal outcomes using insulin detemir or neutral protamine Hagedorn in type 1 diabetes. J Matern Fetal Neonatal Med. 2014 Jan;27(1):7-13. doi: 10.3109/14767058.2013.799650. Epub 2013 Jun 5. PMID 23617228
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted at 79 sites in 17 countries: Denmark, Finland, France, Ireland, United Kingdom, Norway, Croatia, Poland, Austria, Spain, Canada, Argentina, Brazil, South Africa, Russia, Israel and Australia.
Pre-assignment Details: Non-pregnant women were randomised immediately after it was established that they fulfilled the eligibility criteria. Thus, they were exposed to insulin detemir (IDet) throughout organogenesis. Pregnant subjects were to be randomised after completion of the 8th gestational week (GW) and before the completion of 12th GW
Period: Overall Study
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Started | 233 | 237
Exposed-All Subjects | 233 | 232 (5 withdrawn before treatment initiation)
Exposed-Pregnant Subjects | 152 | 158 (3 withdrawn before treatment initiation)
Pregnancies (for Exposed-pregnant) | 152 | 160 (2 subjects had spontaneous abortion and became pregnant again)
Completed | 127 | 136
Not Completed | 106 | 101
Not completed — Adverse Event | 18 | 8
Not completed — Unclassified | 1 | 3
Not completed — Lack of Efficacy | 0 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 10 | 12
Not completed — Withdrawal by Subject | 16 | 18
Not completed — Withdrawal criteria | 60 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin | Total
Number analyzed (Participants) | 152 | 158 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (4.62) | 30.4 (4.21) | 30.1 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 158 | 310
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Black or African American | 1 | 0 | 1
  White | 135 | 142 | 277
  Unknown | 12 | 10 | 22
  Other | 3 | 2 | 5
Height [Mean (Standard Deviation); unit: meters] — The number of subjects (N) analysed in the Neutral Protamine Hagedorn (NPH) group was 157 instead of 158.
  meters | 1.67 (0.07) | 1.65 (0.06) | 1.66 (0.07)
Body Weight [Mean (Standard Deviation); unit: kg] — The number of subjects (N) analysed in the NPH group was 157 instead of 158.
  kg | 67.6 (12.3) | 68.7 (12.4) | 68.2 (12.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The number of subjects (N) analysed in the NPH group was 157 instead of 158.
  kg/m^2 | 24.34 (3.95) | 25.17 (4.22) | 24.76 (4.1)
Smoker [Number; unit: participants]
  No | 143 | 147 | 290
  Yes | 9 | 11 | 20
Daily Use of Alcohol [Number; unit: participants]
  No | 150 | 158 | 308
  Yes | 2 | 0 | 2
Stratification [Number; unit: participants]
  Pregnant after Randomisation | 73 | 75 | 148
  Pregnant at Randomisation | 79 | 83 | 162
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 6.95 (0.82) | 7.08 (0.76) | 7.01 (0.79)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — The number of subjects (N) analysed in the insulin detemir (IDet) group was 139 and NPH group was 151 instead of 152 and 158, respectively.Therefore the total number of subjects analysed were 290 instead of 310.
  mmol/L | 5.89 (3.29) | 5.99 (3.23) | 5.94 (3.25)
Diabetes History [Mean (Standard Deviation); unit: years] | 11.72 (8.08) | 12.78 (7.94) | 12.26 (8.02)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin (HbA1c) for Full Analysis Set (Pregnant Subjects) at GW 36
Time Frame: At gestational week (GW) 36
Population: Full Analysis Set (FAS) for pregnant subjects-all randomised subjects exposed to at least 1 dose of trial drug and pregnant during trial. IDet (N)=152 and NPH (N)=158. Missing values were imputed using Last observation carried forward (LOCF). For FAS, LOCF was made using the pregnancy visits, the early termination visit and the withdrawal visit.
Measure: Least Squares Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 138 | 145
Percent (%) glycosylated haemoglobin | 6.27 (0.053) | 6.33 (0.052)
Statistical Analysis 1: Comparison: Insulin Detemir vs Neutral Protamine Hagedorn (NPH) Insulin; Non-inferiority analysis with a null hypothesis stated that the difference between treatments, IDet-NPH, was equal to or larger than the pre-specified non-inferiority margin of 0.4%. In case non-inferiority was established it was also investigated if IDet was superior to NPH with a null hypothesis stating that the difference between IDet and NPH treatment groups is equal to or greater than 0; Test type: Non-Inferiority or Equivalence — Non-inferiority can only be declared if the non-inferiority criterion was fulfilled for both (FAS and Per-protocol) analysis sets. Non-inferiority was declared if the upper limit of the two-sided 95% CI for the estimated treatment difference was below 0.4%; p = 0.400, Regression, Linear — P-value for superiority was calculated; Treatment, country, pregnancy (preg.) status at randomisation (random.)-fixed. HbA1c at rand.(covariate) & at rand. by preg. status (interaction); Mean Difference (Final Values) = -0.06, 95% CI [-0.21 to 0.08], Standard Error of Mean 0.074 — Estimated treatment differences for IDet versus NPH at Visit P4 with the corresponding 95% confidence interval (CI) was calculated. Non-inferiority was established but superiority was not established

2. Primary Outcome: Glycosylated Haemoglobin (HbA1c) for Per Protocol Analysis Set (Pregnant Subjects) at GW 36
Time Frame: At gestational week (GW) 36
Population: Per Protocol Analysis Set (pregnant subjects): comprised all subjects from the FAS (pregnant subjects) except subjects who significantly violated the inclusion/exclusion criteria. Gestational age at delivery must be at least 32 completed weeks.
Measure: Least Squares Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 127 | 135
Percent (%) glycosylated haemoglobin | 6.22 (0.069) | 6.37 (0.067)
Statistical Analysis 1: Comparison: Insulin Detemir vs Neutral Protamine Hagedorn (NPH) Insulin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.122, Regression, Linear — P-value for superiority was calculated; Treatment, country, preg. status at rand.(fixed factors),HbA1c at rand.(covariate),HbA1c at rand. by preg. status (interaction); Mean Difference (Final Values) = -0.15, 95% CI [-0.34 to 0.04], Standard Error of Mean 0.096 — Estimated treatment differences for IDet versus NPH at Visit P4 with the corresponding 95% CI was calculated. Non-inferiority was established but superiority was not established

3. Secondary Outcome: Glycosylated Haemoglobin (HbA1c) During Pregnancy
Time Frame: During the pregnancy period [Visit P1 (GW 8-12), Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36), Delivery Visit (end of pregnancy)] and Follow-Up Visit ( 6 weeks after delivery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
Percent (%) glycosylated haemoglobin
  GW 8-12 IDet (N)=140, NPH (N)=146 | 6.6 (0.8) | 6.8 (0.7)
  GW 14 IDet (N)=136, NPH (N)=146 | 6.3 (0.7) | 6.5 (0.7)
  GW 24 IDet (N)=138, NPH (N)=146 | 6 (0.7) | 6.1 (0.8)
  GW 36 IDet (N)=138, NPH (N)=146 | 6.2 (0.8) | 6.3 (0.8)
  Delivery IDet (N)=138, NPH (N)=146 | 6.3 (0.7) | 6.5 (1.0)
  Follow-up IDet (N)=138, NPH (N)=146 | 6.5 (0.9) | 6.6 (0.8)

4. Secondary Outcome: Subjects Reaching HbA1c at or Below 6.0% Both at GW 24 and GW 36
Time Frame: At both Visit P3 (GW 24) and Visit P4 (GW 36)
Population: FAS for pregnant subjects-all randomised subjects exposed to at least 1 dose of trial drug and pregnant during trial. IDet (N)=152 and NPH (N)=158. Missing values were imputed using LOCF which was made using pregnancy visits, early termination visit and withdrawal visit. Analysed subjects-subjects with valid HbA1c values at visit P3 and P4.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 138 | 146
participants | 57 | 46

5. Secondary Outcome: Fasting Plasma Glucose (FPG)
Time Frame: During the pregnancy period [Visit P1 (GW 8-12), Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36)]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  GW 8-12 IDet (N)=130, NPH (N)=141 | 5.0 (2.3) | 5.8 (3.0)
  GW 14 IDet (N)=125, NPH (N)=135 | 5.0 (3.0) | 5.7 (2.7)
  GW 24 IDet (N)=129, NPH (N)=141 | 5.2 (2.4) | 6.3 (3.3)
  GW 36 IDet (N)=129, NPH (N)=142 | 4.7 (1.9) | 5.4 (2.3)

6. Secondary Outcome: 8-point Self-monitored Plasma Glucose (SMPG) Profile at GW 24
Description: 8-point SMPG was recorded 3 times prior to each visit, and the average value for each of the 8-time points was applied when presenting and analysing the SMPG data. Visit reallocation was made for the early termination visit and for the withdrawal visit.
Time Frame: Visit P3 (GW 24)
Population: Full Analysis Set (FAS) for pregnant subjects-all randomised subjects exposed to at least 1 dose of trial drug and pregnant during trial. IDet (N)=152 & NPH (N)=158. Missing values were imputed using Last observation carried forward (LOCF). For FAS, LOCF was made using the average values.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  Before Breakfast (N=131,141) | 6.4 (1.9) | 7.3 (2.0)
  120 mins after breakfast (N=130,141) | 7.7 (2.3) | 8.0 (2.2)
  Before Lunch (N=131,141) | 6.1 (1.9) | 6.7 (2.1)
  120 mins after lunch (N=130,140) | 7.2 (1.9) | 7.4 (2.1)
  Before Dinner (N=130,140) | 6.8 (2.0) | 7.0 (2.1)
  120 mins after Dinner (N=117,133) | 7.2 (2.0) | 7.8 (2.1)
  Bedtime (N=125,137) | 7.6 (2.4) | 7.8 (2.2)
  At 2.00 A.M. (N=125,134) | 6.7 (2.1) | 6.9 (2.3)

7. Secondary Outcome: 8-point Self Monitored Plasma Glucose (SMPG) Profile at GW 36
Description: as for outcome 6
Time Frame: Visit P4 (GW 36)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  Before Breakfast (N=131,141) | 6 (1.7) | 6.3 (1.6)
  120 mins after breakfast (N=130,139) | 7.4 (2) | 7.5 (1.9)
  Before Lunch (N=131,141) | 5.9 (1.7) | 6.1 (1.9)
  120 mins after lunch (N=130,140) | 6.9 (1.7) | 7.1 (2.1)
  Before Dinner (N=131,140) | 6.5 (1.7) | 6.5 (1.9)
  120 mins after Dinner (N=117,132) | 7.4 (2.1) | 7.4 (1.9)
  Bedtime (N=126,137) | 7 (1.8) | 7.2 (2)
  At 2.00 A.M. (N=122,135) | 6 (1.8) | 6.4 (1.8)

8. Secondary Outcome: Maternal Safety - Number of Subjects With Adverse Events (AEs)
Description: AE=any undesirable medical event occurring to a subject in a clinical trial, whether or not related to the trial product. Related AE=relationship of probable or possible. Serious adverse event (SAE) =any undesirable serious medical event as defined in protocol.
Time Frame: Participants were followed during the pregnancy period, an average of 9.6 months
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
participants
  Subjects with (w.) adverse events | 138 | 141
  Subjects with serious adverse events | 61 | 49
  Subjects with severe adverse events | 38 | 32
  Subjects w. AEs related to basal insulin | 18 | 16
  Subjects w. AEs related to bolus insulin | 12 | 14
  Subjects with AEs leading to withdrawal | 13 | 6

9. Secondary Outcome: Safety in Children - Number of Subjects (Foetuses and Newborns) With Adverse Events
Description: AE=any undesirable medical event occurring to a subject in a clinical trial, whether or not related to the trial product. Related AE=relationship of probable or possible. SAE=any undesirable serious medical event as defined in protocol.
Time Frame: Foetuses/Newborns were followed during the pregnancy period, an average of 9.6 months and Follow-Up period (6 weeks after delivery)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. Each pregnant woman analyzed had exactly one Foetus/Newborn that was analyzed for AEs.
Measure: Number; unit: Foetus/Newborns (1 per pregnant woman)
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
Foetus/Newborns (1 per pregnant woman)
  Subjects with adverse events | 56 | 55
  Subjects with serious adverse events | 36 | 32
  Subjects with severe adverse events | 15 | 12
  Subjects w. AEs related to Basal insulin | 1 | 0
  Subjects w. AEs related to Bolus insulin | 1 | 0
  Subjects with AEs leading to withdrawal | 0 | 1

10. Secondary Outcome: Maternal Safety - Hypoglycaemic Episodes
Description: All episodes include major, minor and symptoms only. Major episode : unable to self-treat. Minor: able to self-treat and plasma glucose (PG) < 3.1 mmol/L. Symptoms only: able to self-treat and no PG measurement or PG glucose ≥3.1 mmol/L. Diurnal: Episode occurring between 06.00 - 00.00, both including.
Time Frame: Participants were followed during the pregnancy period, an average of 9.6 months
Population: as for outcome 8
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 144 | 146
episodes
  All Episodes | 9496 | 9453
  Diurnal | 8045 | 7810

11. Secondary Outcome: Maternal Safety - Nocturnal Hypoglycaemic Episodes
Description: A nocturnal episode is any episode occurring between 0.01 - 5.59, both including. It includes major, minor and symptoms only episodes. Major: unable to self-treat. Minor: able to self-treat and plasma glucose (PG) < 3.1 mmol/L. Symptoms only: able to self-treat and no PG measurement or PG glucose ≥3.1 mmol/L.
Time Frame: Participants were followed during the pregnancy period, an average of 9.6 months
Population: as for outcome 8
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 119 | 130
episodes | 1451 | 1643

12. Secondary Outcome: Maternal Safety - Change in Albumin Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in albumin level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
g/dL
  Visit P1 IDet (N)=138, NPH (N)=145 | 4.05 (0.22) | 4.04 (0.23)
  FU Visit IDet (N)=138, NPH (N)=146 | 4.19 (0.25) | 4.12 (0.27)
  Change from Visit P1-FU (N=136, 145) | 0.13 (0.26) | 0.09 (0.26)

13. Secondary Outcome: Maternal Safety - Change in Alanine Aminotransferase Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in alanine aminotransferase level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
U/L
  Visit P1 IDet (N)=138, NPH (N)=145 | 16.12 (11.31) | 17.97 (9.53)
  FU Visit IDet (N)=138, NPH (N)=146 | 27.06 (14.92) | 26.16 (14.21)
  Change from Visit P1-FU (N=136, 145) | 10.88 (17.51) | 8.16 (15.6)

14. Secondary Outcome: Maternal Safety - Change in Alkaline Phosphatase Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in alkaline phosphatase level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
U/L
  Visit P1 IDet (N)=137, NPH (N)=144 | 52.64 (13.63) | 53.88 (13.75)
  FU Visit IDet (N)=138, NPH (N)=146 | 90.17 (26.68) | 92.96 (28.07)
  Change from Visit P1-FU (N=135, 144) | 37.39 (20.86) | 39.51 (23.34)

15. Secondary Outcome: Maternal Safety - Change in Creatinine Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in creatinine serum level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mcmol/L
  Visit P1 IDet (N)=138, NPH (N)=145 | 52.04 (7.85) | 54.01 (8.81)
  FU Visit IDet (N)=138, NPH (N)=146 | 62.98 (9.73) | 66.57 (11.8)
  Change from Visit P1-FU (N=136, 145) | 11.18 (7.61) | 12.52 (8.67)

16. Secondary Outcome: Maternal Safety - Change in Lactate Dehydrogenase Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in lactate dehydrogenase serum level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
U/L
  Visit P1 IDet (N)=138, NPH (N)=145 | 145.1 (34.11) | 144.1 (24.6)
  FU Visit IDet (N)=138, NPH (N)=146 | 167.5 (29.29) | 169.5 (33.75)
  Change from Visit P1-FU (N=136, 145) | 21.82 (33.61) | 25.46 (30.48)

17. Secondary Outcome: Maternal Safety - Change in Potassium Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in potassium serum level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  Visit P1 IDet (N)=137, NPH (N)=144 | 4.13 (0.32) | 4.12 (0.27)
  FU Visit IDet (N)=138, NPH (N)=146 | 4.30 (0.33) | 4.31 (0.34)
  Change from Visit P1-FU (N=135, 144) | 0.15 (0.36) | 0.20 (0.36)

18. Secondary Outcome: Maternal Safety - Change in Sodium Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in sodium serum level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  Visit P1 IDet (N)=137, NPH (N)=145 | 138.0 (2.19) | 137.8 (2.36)
  FU Visit IDet (N)=138, NPH (N)=146 | 141.6 (2.57) | 141.2 (2.71)
  Change from Visit P1-FU (N=135, 145) | 3.59 (3.19) | 3.36 (3.27)

19. Secondary Outcome: Maternal Safety - Change in Total Protein Serum Level (Biochemistry)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in total protein serum level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial.Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
g/dL
  Visit P1 IDet (N)=138, NPH (N)=145 | 6.84 (0.37) | 6.89 (0.42)
  FU Visit IDet (N)=138, NPH (N)=146 | 7.08 (0.44) | 7.11 (0.47)
  Change from Visit P1-FU (N=136, 145) | 0.24 (0.42) | 0.22 (0.39)

20. Secondary Outcome: Maternal Safety - Change in Haemoglobin Level (Haematology)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in haemoglobin level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmol/L
  Visit P1 IDet (N)=138, NPH (N)=146 | 7.64 (0.48) | 7.64 (0.5)
  FU Visit IDet (N)=138, NPH (N)=146 | 7.81 (0.57) | 7.69 (0.57)
  Change from Visit P1-FU (N=136, 145) | 0.16 (0.57) | 0.05 (0.6)

21. Secondary Outcome: Maternal Safety - Change in Leukocytes Level (Haematology)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in leukocytes level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
10^9 cells/L
  Visit P1 IDet (N)=138, NPH (N)=146 | 8.01 (2.21) | 8.2 (2.04)
  FU Visit IDet (N)=138, NPH (N)=146 | 6.68 (1.79) | 6.55 (1.92)
  Change from Visit P1-FU (N=136, 145) | -1.36 (1.93) | -1.65 (2.12)

22. Secondary Outcome: Maternal Safety - Change in Thrombocytes Level (Haematology)
Description: This is the standard safety lab parameter and is calculated as an estimate of the mean change from Visit P1 in thrombocytes level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
10^9 cells/L
  Visit P1 IDet (N)=138, NPH (N)=146 | 245.3 (48.27) | 247.2 (59.32)
  FU Visit IDet (N)=138, NPH (N)=146 | 270.6 (66.01) | 263.1 (68.12)
  Change from Visit P1-FU (N=136, 145) | 24.25 (55.07) | 16.16 (52.02)

23. Secondary Outcome: Maternal Safety - Change in Urine Albumin Level (Urinalysis)
Description: This is the standard safety lab parameter and calculated as an estimate of the mean change from Visit P1 in urine albumin level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
g/dL
  Visit P1 IDet (N)=135, NPH (N)=143 | 0.01 (0.02) | 0.01 (0.02)
  FU Visit IDet (N)=138, NPH (N)=146 | 0.02 (0.04) | 0.03 (0.12)
  Change from Visit P1-FU (N=133, 142) | 0.01 (0.04) | 0.02 (0.11)

24. Secondary Outcome: Maternal Safety - Change in Albumin/Creatinine Ratio (Urinalysis)
Description: This is the standard safety lab parameter and calculated as an estimate of the mean change from Visit P1 in albumin/creatinine ratio at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mg/mmol
  Visit P1 IDet (N)=135, NPH (N)=143 | 0.82 (1.4) | 0.85 (1.65)
  FU Visit IDet (N)=138, NPH (N)=146 | 2.65 (5.6) | 4.81 (32.22)
  Change from Visit P1-FU (N=133, 142) | 1.88 (5.29) | 4.07 (32.43)

25. Secondary Outcome: Maternal Safety - Change in Urine N (Creatinine) (Urinalysis)
Description: This is the standard safety lab parameter and calculated as an estimate of the mean change from Visit P1 in Urine-N (creatinine) level at Follow-Up Visit (6 weeks after delivery).
Time Frame: Visit P1 (GW 8-12), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mg/dL
  Visit P1 IDet (N)=135, NPH (N)=144 | 114.8 (63.77) | 103.1 (56.37)
  FU Visit IDet (N)=138, NPH (N)=146 | 106.2 (66.44) | 98.61 (58.71)
  Change from Visit P1-FU (N=133, 143) | -6.62 (83.83) | -6.34 (70.79)

26. Secondary Outcome: Maternal Safety - Change in Insulin Detemir Specific Antibodies
Description: Change in concentrations of values for insulin detemir specific antibodies from baseline to Visit P4 was calculated. The unit for measuring antibody levels is amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture (%B/T). Samples were taken before 1st dosing.
Time Frame: Baseline, Visit P4 (GW 36). Baseline is Visit 2 (randomisation visit, within 3 weeks of screening) for subjects not pregnant at randomisation and Visit P1 (GW 8-12) for pregnant subjects at randomisation.
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
%B/T
  Baseline IDet (N)=145, NPH (N)=155 | 1.13 [-0.10 to 6.55] | 1.09 [-1.36 to 7.35]
  Visit P4 IDet (N)=110, NPH (N)=110 | 1.36 [-0.64 to 12.71] | 1.25 [-3.64 to 6.74]
  Change from Baseline-Visit P4(N=105,109) | 0.04 [-3.89 to 12.11] | 0.09 [-5.93 to 6.26]

27. Secondary Outcome: Maternal Safety - Change in Insulin Aspart Specific Antibodies
Description: Change in concentrations values for insulin aspart specific antibodies from baseline to Visit P4 was calculated. The unit for measuring antibody levels is amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture (%B/T). Samples were taken before 1st dosing.
Time Frame: as for outcome 26
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
%B/T
  Baseline IDet (N)=145, NPH (N)=154 | 0.44 [-0.25 to 29.74] | 0.46 [-0.39 to 55.73]
  Visit P4 IDet (N)=109, NPH (N)=110 | 0.43 [-0.58 to 22.34] | 0.36 [-0.52 to 52.23]
  Change from Baseline-Visit P4(N=104,109) | -0.12 [-8.63 to 10.10] | -0.21 [-11.6 to 2.11]

28. Secondary Outcome: Maternal Safety - Change in Insulin Detemir/Insulin Aspart Cross Reacting Antibodies
Description: Change in concentrations values for insulin detemir/aspart cross-reacting antibodies from baseline to Visit P4 was calculated. The unit for measuring antibody levels is amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture (%B/T). Samples were taken before 1st dosing
Time Frame: as for outcome 26
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
%B/T
  Baseline IDet (N)=146, NPH (N)=155 | 5.21 [-0.02 to 76.75] | 5.36 [-0.50 to 67.4]
  Visit P4 IDet (N)=110, NPH (N)=110 | 5.40 [-0.21 to 50.37] | 4.28 [-0.22 to 62.25]
  Change from Baseline-Visit P4(N=106,109) | -0.43 [-43.3 to 39.43] | -1.12 [-27.9 to 14.52]

29. Secondary Outcome: Pregnancy Outcome Safety - Level of Detemir Specific Antibodies (AB) in Umbilical Cord Blood
Description: Antibodies were measured in a subtraction radioimmunoassay and expressed as antibody bound tracer relative to the total amount of tracer (%B/T).
Time Frame: At Delivery (End of Pregnancy)
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 104 | 118
%B/T | 1.31 [-0.43 to 13.74] | 0.90 [-2.48 to 3.23]

30. Secondary Outcome: Pregnancy Outcome Safety - Level of Aspart Specific Antibodies (AB) in Umbilical Cord Blood
Description: as for outcome 29
Time Frame: At Delivery (End of Pregnancy)
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 103 | 118
%B/T | 0.38 [-0.87 to 19.27] | 0.32 [-0.45 to 11.08]

31. Secondary Outcome: Pregnancy Outcome Safety - Level of Cross-Reacting Antibodies (AB) in Umbilical Cord Blood
Description: as for outcome 29
Time Frame: At Delivery (End of Pregnancy)
Population: as for outcome 8
Measure: Median (Full Range); unit: %B/T
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 104 | 119
%B/T | 5.99 [0.06 to 49.67] | 4.12 [0.05 to 74.59]

32. Secondary Outcome: Ratio Between Detemir Specific Antibodies in Cord Blood and Maternal Antibodies
Description: Cord blood (at delivery) vs. Maternal Blood at Visit P4 (GW 36)
Time Frame: At Delivery (End of Pregnancy) and at Visit P4 (GW 36)
Population: as for outcome 8
Measure: Median (Full Range); unit: ratio
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 94 | 96
ratio | 1.10 [-39.2 to 8.80] | 0.77 [-4.20 to 7.50]

33. Secondary Outcome: Pregnancy Outcome Safety - Level of Insulin Detemir in Umbilical Cord Blood
Time Frame: At Delivery
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. IDet in cord blood was analysed for subjects in the IDet Arm and only for 98 subjects, as for 72 subjects it was reported as below measuring range (<25.00 pmol/L).
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 98 | 0
pmol/L | 25.00 [25.00 to 209.6] |

34. Secondary Outcome: Maternal Safety - Change From Visit P1 in Body Weight During Pregnancy by Visit
Description: Change in the body weight was summarised by treatment.
Time Frame: Visit P1 (GW (8-12), Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. Missing values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
kg
  GW (8-12) IDet(N)=139,NPH(N)=145 | 67.8 (11.6) | 69.2 (12.5)
  Change from GW(8-12)-GW 14 (N=128,139) | 1.0 (1.6) | 1.4 (1.9)
  Change from GW(8-12)-GW 24 (N=130,139) | 5.6 (2.7) | 6.0 (3.2)
  Change from GW(8-12)-GW 36(N=130,139) | 11.5 (4.2) | 11.0 (5.2)

35. Secondary Outcome: Maternal Safety - Change From Visit P1 in Systolic Blood Pressure During Pregnancy and at Follow-Up by Visit
Description: Change in the systolic blood pressure was summarised by treatment.
Time Frame: Visit P1 (GW (8-12)), Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36), Follow-Up (FU) Visit (6 weeks after delivery)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmHg
  GW (8-12) IDet(N)=140,NPH(N)=146 | 114.1 (11.4) | 116.2 (10.4)
  Change from GW(8-12)-GW 14 (N=137,145) | 0.8 (10.1) | -2.8 (9.6)
  Change from GW(8-12)-GW 24(N=138,145) | -0.7 (9.6) | -1.6 (11.3)
  Change from GW(8-12)-GW 36(N=138,145) | 3.1 (11.3) | 2.3 (11.8)
  Change from GW(8-12)-FU(N=138,145) | 2.6 (11.6) | -0 (12.5)

36. Secondary Outcome: Maternal Safety - Change From Visit P1 in Diastolic Blood Pressure During Pregnancy and at Follow-Up by Visit
Description: Change in the diastolic blood pressure was summarised by treatment.
Time Frame: as for outcome 35
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
mmHg
  GW (8-12) IDet(N)=140,NPH(N)=146 | 70.5 (8.9) | 70.7 (8.2)
  Change from GW(8-12)-GW 14 (N=137,145) | -0.2 (8.4) | -0.5 (9.1)
  Change from GW(8-12)-GW 24(N=138,145) | -1.6 (8.7) | -1.2 (9.3)
  Change from GW(8-12)-GW 36(N=138,145) | 3.2 (9.9) | 2.6 (11.0)
  Change from GW(8-12)-FU(N=138,145) | 1.3 (9.5) | 1.8 (9.8)

37. Secondary Outcome: Maternal Safety - Change From Visit P1 in Pulse During Pregnancy and at Follow-Up
Description: Change in the pulse was summarised by treatment.
Time Frame: Visit P1 (GW (8-12), Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36), Follow-Up Visit (6 weeks after delivery)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
beats/minute
  GW (8-12) IDet(N)=136,NPH(N)=142 | 77.4 (10) | 76.8 (9.6)
  Change from GW(8-12)-GW 14 (N=133,139) | 1.5 (9.3) | 2.2 (10)
  Change from GW(8-12)-GW 24(N=134,141) | 3.5 (10.6) | 4.5 (10.6)
  Change from GW(8-12)-GW 36(N=134,141) | 5.2 (11.8) | 4.9 (12)
  Change from GW(8-12)-FU(N=134,141) | -3 (11.7) | -2.3 (11.9)

38. Secondary Outcome: Maternal Safety - Electrocardiogram (ECG)
Description: The number of subjects having a electrocardiogram (ECG) that changed from 'Normal' or 'Abnormal, not clinically significant' (at Visit 1, 3 weeks before randomisation) to 'Abnormal, clinically significant' (at Follow-Up). 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Follow-Up (6 weeks after delivery)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
participants | 0 | 0

39. Secondary Outcome: Maternal Safety - Acceleration of Retinopathy in Any Eye
Description: Acceleration of Retinopathy is defined as worsening of fundoscopy/fundusphotography findings from GW 8-12 (Visit P1) to follow-up on one or both eyes.
Time Frame: From GW 8-12 (Visit P1) to Follow-Up (6 weeks after delivery)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. Acceleration of retinopathy was summarised by treatment and missing data was imputed using LOCF.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
participants
  Acceleration in Any Eye | 12 | 14
  No Acceleration in Any Eye | 120 | 120
  Missing Data | 20 | 24

40. Secondary Outcome: Maternal Safety - Acceleration of Nephropathy
Description: Acceleration of nephropathy was defined as a change from a low U-albumin:U-creatinine ratio ≤33.93 mg/mmol to a high U-albumin:U-creatinine ratio > 33.93 mg/mmol from GW 8-12 (Visit P1) to the follow-up visit.
Time Frame: From GW 8-12 (Visit P1) to Follow-Up (6 weeks after delivery)
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. Acceleration of nephropathy was summarised by treatment and missing data was imputed using LOCF.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
participants | 2 | 1

41. Secondary Outcome: Maternal Safety - Mode of Delivery
Description: Non-Planned Caesarean Section is a procedure which takes place ≤8h prior to delivery. Planned Caesarean Section takes place >8h prior to delivery.
Time Frame: At Delivery Visit
Population: Safety analysis set (pregnant subjects): all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial. This set in total contains 152 subjects in IDet and 158 subjects in NPH arm. The partcipant analysed for this outcome measure are the number of subjects at delivery visit.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 130 | 136
percentage (%) of subjects
  Spontaneous onset of labour (N)=130,136 | 19 | 28
  Induction of labour (N)=130,136 | 39 | 36
  Normal Vaginal Delivery(N)=54,50 | 76 | 80
  Instrumental Vaginal Delivery(N)=54,50 | 24 | 20
  Non-Planned Caesarean Section(N)=76,86 | 36 | 43
  Planned Caesarean Section(N)=76,86 | 65 | 57

42. Secondary Outcome: Pregnancy Outcome at Delivery
Description: Induced abortion means interruption of a living pregnancy < 22 completed weeks. Early foetal death means death before 22 completed GWs. Stillbirth indicates death between at or after 22 GW and at or before delivery.
Time Frame: Delivery Visit
Population: Safety analysis set (pregnant subjects): randomised subjects exposed to at least 1 dose of trial product and preg. during the trial. IDet (N)=152 (152 pregnancies) NPH (N)=158 subjects (160 pregnancies, 2 subjects had spontaneous abortion and became preg. again). Analysed subjects-no. of subjects with a preg. outcome at delivery visit.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 142 | 145
participants
  Live Birth | 128 | 136
  Early Foetal Death (Spont. Abortion) | 10 | 8
  Early Foetal Death (Ectopic Pregnancy) | 1 | 1
  Induced Abortion | 1 | 0
  Stillbirth | 2 | 0

43. Secondary Outcome: Pregnancy Outcome at Follow-Up
Description: Induced abortion means interruption of a living pregnancy < 22 completed weeks. Early foetal death means death before 22 completed GWs. Perinatal Death means death of a foetus/infant between ≥ 22 completed GWs and < 1 completed week after delivery. Neonatal Death means death between at or after 7 completed days and before 28 completed days after delivery. Death During Follow-Up means death between at or after 28 days after delivery and at or before Follow-Up.
Time Frame: Follow-Up (6 weeks after delivery)
Population: as for outcome 42
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 142 | 145
participants
  Live Children | 128 | 135
  Early Foetal Death (Spont. Abortion) | 10 | 8
  Early Foetal Death (Ectopic Pregnancy) | 1 | 1
  Induced Abortion | 1 | 0
  Perinatal Death | 2 | 1
  Neonatal Death | 0 | 0
  Death During Follow-Up | 0 | 0

44. Secondary Outcome: Safety - Total Daily Insulin Dose During Pregnancy
Time Frame: Visit P2 (GW 14), Visit P3 (GW 24), Visit P4 (GW 36), Follow-Up (6 weeks after delivery)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
U/kg
  GW 14 IDet (N)=129, NPH (N)=141 | 0.73 (0.23) | 0.74 (0.25)
  GW 24 IDet (N)=128, NPH (N)=137 | 0.85 (0.29) | 0.84 (0.26)
  GW 36 IDet (N)=119, NPH (N)=121 | 1.17 (0.47) | 1.05 (0.35)
  Follow-Up IDet (N)=124, NPH (N)=133 | 0.53 (0.17) | 0.57 (0.2)

45. Secondary Outcome: Safety - Composite Pregnancy Outcome
Description: Wt. corresponds to weight of live-born infants. Pre-term delivery: delivery before 37 completed GWs including abortions. Early foetal death: death before 22 completed GWs. Perinatal mortality: death of a foetus/infant between ≥ 22 completed GWs and < 1 completed week after delivery. Neonatal mortality: post-partum after 7 completed days and before 28 completed days after delivery. Major-malformation: a life threatening structural anomaly or one likely to cause significant impairment of health or functional capacity and needs medical or surgical treatment.
Time Frame: End of Pregnancy
Population: Safety analysis set (pregnant subjects): randomised subjects exposed to at least 1 dose of trial product and pregnant during the trial. IDet (N)=152 (152 pregnancies) NPH (N)=158 subjects (160 pregnancies, 2 subjects had spontaneous abortion and became pregnant again).
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 152 | 158
participants
  Wt. below the 10th percentile(N)=128,136 | 3 | 1
  Wt. above the 90th percentile(N)=128,136 | 59 | 73
  Pre-term delivery (N)=142,145 | 39 | 45
  Major malformations (N)=142,145 | 5 | 1
  Early foetal death (N)=142,145 | 11 | 9
  Perinatal mortality (N)=130,136 | 2 | 1
  Neonatal mortality (N)=126,135 | 0 | 0
  Compiled(at least 1 of above)(N)=142,145 | 89 | 96

46. Secondary Outcome: Ratio Between Aspart Specific Antibodies in Cord Blood and Maternal Antibodies
Description: Cord blood (at delivery) vs. Maternal Blood at Visit P4 (GW 36)
Time Frame: At Delivery (End of Pregnancy) and at Visit P4 (GW 36)
Population: as for outcome 8
Measure: Median (Full Range); unit: ratio
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 93 | 95
ratio | 0.84 [-2.85 to 8.0] | 0.64 [-25.5 to 5.0]

47. Secondary Outcome: Ratio Between Cross-reacting Antibodies in Cord Blood and Maternal Antibodies
Description: Cord blood (at delivery) vs. Maternal Blood at Visit P4 (GW 36)
Time Frame: At Delivery (End of Pregnancy) and at Visit P4 (GW 36)
Population: as for outcome 8
Measure: Median (Full Range); unit: ratio
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Number analyzed (Participants) | 94 | 98
ratio | 1.29 [-76.0 to 8.83] | 0.90 [-3.86 to 57.82]

ADVERSE EVENTS:
Time Frame: Maternal AEs were collected and reported during the entire pregnancy period, an average of 9.6 months
Description: AEs has been reported for Mother (during the pregnancy) in the safety analysis set for pregnant subjects (Safety-Pregnant) comprising of all randomised subjects who were exposed to at least one dose of trial product and who were pregnant during the trial.
Arm/Group | Insulin Detemir | Neutral Protamine Hagedorn (NPH) Insulin
Serious Adverse Events (participants affected / at risk) | 61/152 | 49/158
Other Adverse Events (participants affected / at risk) | 138/152 | 141/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=152) | Neutral Protamine Hagedorn (NPH) Insulin (N=158)
Aborption spontaneous (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 4 (4) — SAE for Mother, Safety-Pregnant
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 1 (1) — SAE for Mother, Safety-Pregnant
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) — SAE for Mother, Safety-Pregnant
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) — SAE for Mother, Safety-Pregnant
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) — SAE for Mother, Safety-Pregnant
Abortion threatened (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — SAE for Mother, Safety-Pregnant
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) — SAE for Mother, Safety-Pregnant
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — SAE for Mother, Safety-Pregnant
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — SAE for Mother, Safety-Pregnant
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — SAE for Mother, Safety-Pregnant
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — SAE for Mother, Safety-Pregnant
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2) — SAE for Mother, Safety-Pregnant
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) — SAE for Mother, Safety-Pregnant
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — SAE for Mother, Safety-Pregnant
Aborption incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Antepartum haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Labour complication (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Placental insufficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (12) — SAE for Mother, Safety-Pregnant
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 2 (4) | 7 (9) — SAE for Mother, Safety-Pregnant
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 (5) | 1 (1) — SAE for Mother, Safety-Pregnant
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) — SAE for Mother, Safety-Pregnant
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — SAE for Mother, Safety-Pregnant
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) — SAE for Mother, Safety-Pregnant
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) — SAE for Mother, Safety-Pregnant
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 1 (2) — SAE for Mother, Safety-Pregnant
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) — SAE for Mother, Safety-Pregnant
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1) — SAE for Mother, Safety-Pregnant
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Urogenital infection bacterial (Infections and infestations) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2) — SAE for Mother, Safety-Pregnant
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) — SAE for Mother, Safety-Pregnant
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Headache (Nervous system disorders) | 3 (3) | 2 (2) — SAE for Mother, Safety-Pregnant
Migraine (Nervous system disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — SAE for Mother, Safety-Pregnant
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Hypertension (Vascular disorders) | 2 (3) | 1 (1) — SAE for Mother, Safety-Pregnant
Retinopathy (Eye disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Visual impairment (Eye disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Device failure (General disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Malaise (General disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Cytolytic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Inadequate diet (Social circumstances) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Social stay hospitalisation (Social circumstances) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
Amniotic fluid volume decreased (Investigations) | 1 (1) | 0 (0) — SAE for Mother, Safety-Pregnant
Polymorphic eruption of pregnancy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — SAE for Mother, Safety-Pregnant
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=152) | Neutral Protamine Hagedorn (NPH) Insulin (N=158)
Nasopharyngitis (Infections and infestations) | 45 (82) | 47 (68) — AE for Mother, Safety-Pregnant
Urinary Tract Infection (Infections and infestations) | 17 (19) | 12 (14) — AE for Mother, Safety-Pregnant
Gastroenteritis (Infections and infestations) | 13 (13) | 9 (11) — AE for Mother, Safety-Pregnant
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 13 (17) — AE for Mother, Safety-Pregnant
Influenza (Infections and infestations) | 9 (12) | 16 (16) — AE for Mother, Safety-Pregnant
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 10 (10) — AE for Mother, Safety-Pregnant
Headache (Nervous system disorders) | 43 (109) | 35 (121) — AE for Mother, Safety-Pregnant
Diarrhoea (Gastrointestinal disorders) | 21 (27) | 11 (13) — AE for Mother, Safety-Pregnant
Abdominal Pain (Gastrointestinal disorders) | 11 (15) | 12 (22) — AE for Mother, Safety-Pregnant
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 5 (7) — AE for Mother, Safety-Pregnant
Toothache (Gastrointestinal disorders) | 7 (9) | 9 (12) — AE for Mother, Safety-Pregnant
Constipation (Gastrointestinal disorders) | 4 (4) | 11 (11) — AE for Mother, Safety-Pregnant
Diabetic Retinopathy (Eye disorders) | 6 (6) | 10 (13) — AE for Mother, Safety-Pregnant
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 13 (17) — AE for Mother, Safety-Pregnant
Anaemia (Blood and lymphatic system disorders) | 22 (23) | 23 (24) — AE for Mother, Safety-Pregnant
Hypertension (Vascular disorders) | 5 (5) | 8 (8) — AE for Mother, Safety-Pregnant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk (NN) reserves the right not to release data until specified milestones, e.g. Clinical Trial Report is available. This includes the right not to release interim results, because the release of such information can invalidate the results of the trial. At the end of the trial, one or more manuscripts for publication will be prepared in collaboration between authors and NN. NN reserves the right to postpone publication and communication for a short time to protect intellectual property.